CLINICAL TRIAL: NCT03077425
Title: Obesity and Caries in Young South Asian Children: A Common Risk Factor Approach
Acronym: CHALO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Columbia University (Other); Rutgers University (Other); University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-6156
Record Dates: First submitted 2017-03-02; First posted 2017-03-13 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Pediatric Obesity; Early Childhood Caries
MeSH Terms: conditions — Pediatric Obesity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Research Assessment- at 6, 12, and 18 months will be conducted by RAs. Data collected include a computerized 24 hour recall: MySmileBuddy (see below); and questionnaires. The T2 interview, in addition, will include the Intra-oral Camera Caries Assessment. Study identifiers will not include indication of group assignment. The REDCap database will include group assignment in a field that is not accessible to RAs
  Caries Outcomes- Intra-oral camera images will be transmitted electronically to the University of Rochester; no group assignment identifier will be included.
  Obesity Outcomes- RAs will obtained weight and length measures in the home- see above.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): An RCT will enroll 360 mothers (total) of children 4-6 month olds from New York City (n=3) and New Jersey (n=2) pediatric practices. Half (180) will be assigned to the Community Health Worker intervention comprised of: a) home visits with mothers/families (n=6 visits over one year) and follow up telephone support; b) patient navigation to make/keep timely dental visits (2x by 18 months).
  Interventions: Behavioral: Intervention
- Enhanced Usual Care (EUC) (Placebo Comparator): Community Health Workers (CHWs)- will deliver the EUC to all study participants at their 6 month well-child visit, which will occur just after their T0 Baseline Interview, just prior to randomization. EUC Components: 1) Pamphlet- CHWs will hand out and review deliver and review a pamphlet with basic ECC and Obesity prevention messages for parents of 6-18 month olds; and 2) Dental Referral List of dentists who will see 12 month olds, and who accept most insurance plans in the pediatric practices we are recruiting from.
  Thus, the EUC will be delivered to n=180 families in the EUC Control and n=180 families in the Intervention group.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Enhanced Usual Care (EUC) — Per Arm/Group Description, CHWs will provide a pamphlet and dental referral list to participants both groups.
  Arms: Enhanced Usual Care (EUC)
Behavioral: Intervention — Per Arm/Group Description, CHWs will a) conduct 6 home visits with mothers/families over a 12 month period along with follow-up phone support, and b) patient navigation support for child to receive 2 dental visits: one by 12 months of age and one by 18 months of age.
  Arms: Intervention

SUMMARY:
The CHALO ("Child Health Action to Lower Oral Caries and Obesity") -- from an Urdu word meaning "Let's go!"-is a multi-level strategy to reduce pediatric obesity and dental caries risk in South Asian (SA) children. Obesity and caries are the two most prominent health disparities of early childhood. Both caries and obesity: a) disproportionately impact low-income children of color, b) share common risk behaviors, i.e., feeding practices, and c) can most effectively be reduced or prevented prevention in infancy and early childhood. SA immigrant children are at high risk for both. CHALO includes both a randomized controlled trial (RCT) aimed at reducing risk behavior, and a Knowledge Translation project to raise awareness in SA lay and professional communities regarding child health risks.

DETAILED DESCRIPTION:
CHALO builds upon the team's prior research re: cariogenic (R34-DE-022282) and obesogenic behaviors (10, 14, 15). CHALO's intervention components-- home visits, phone support, and "patient navigation" to dental visits-- proved to be feasible and acceptable. In the pilot R34, there were promising behavioral change on all measures. CHALO builds on this work, with the addition of: a) sippy cups as an intervention target, b) an iPad-based dietary recall tool, "MySmileBuddy," c) caries and obesity data, and; d) increased intervention contacts- consistent with recent child obesity and caries interventions (16, 17).

An RCT (Aim 1) will enroll 360 mothers of children 4-6 month olds from New York City (n=3) and New Jersey (n=2) pediatric practices in SAPPHIRE ("SA Practice Partnership for Health Improvement and Research"). The Community Health Worker intervention includes: a) home visits with mothers/families (n=6 visits over one year) and follow up telephone support; b) patient navigation to make/keep timely dental visits (2x by 18 months). The Knowledge Translation component (Aim 2) will raise awareness of child health risks in SA communities and among professionals who provide their care. The campaign will include both traditional and social media components and will be evaluated using multiple metrics.

ELIGIBILITY:
Inclusion Criteria:

* Age: Child is < 6 months of age at time of recruitment
* Insurance: Child is enrolled in either Medicaid or CHIP
* Nativity- Mother was born in India, Pakistan, or Bangladesh)
* Language- Mother speaks standard Bengali, English or Hindi/Urdu
* Agency- Mother is index child's primary caretaker.

Exclusion Criteria:

* Inability to provide informed consent per RA judgment
* Plans to travel for > 1 month during follow-up, and
* child health condition barring participation (per pediatrician review of recruitment lists).

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 380 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Quantity of (Combined) Sippy Cup and/or Bottles (Common Risk/Behavioral) | 18 months of age (final follow-up [T2])
  Number and amount of sippy cups + bottles/day consumed by child, obtained by RA assessment using MySmileBuddy

SECONDARY OUTCOMES:
Added Sweeteners/Solids (Common Risk/Behavioral) | 18 months of age (final follow-up [T2])
  Number of sweeteners and/or solids/day added to child's sippy sups/bottles, obtained by RA
Fruits & Vegetables (Common Risk/Behavioral) | 18 months of age (final follow-up [T2])
  Frequency of servings/day obtained by RA assessment using MySmileBuddy
Juice & Sweet Drinks (Common Risk/Behavioral) | 18 months of age (final follow-up [T2])
  Frequency of servings/day obtained by RA assessment using MySmileBuddy
Use of Bottles/Sippy Cups at Nap or Bedtime (Common Risk/Behavioral) | 18 months of age (final follow-up [T2])
  Frequency of child drinking from a bottle or sippy cup/day when put down to bed or nap by RA assessment using MySmileBuddy
Sweet & Salty Snacks (Common Risk/Behavioral) | 18 months of age (final follow-up [T2])
  Frequency of servings obtained by RA assessment using MySmileBuddy
Physical Activity (Obesity/Behavioral) | 18 months of age (final follow-up [T2])
  Time child spent in active play, assessed by parent completed questionnaire
Screen Time (Obesity/Behavioral) | 18 months of age (final follow-up [T2])
  Time child spent in front of TV, computer, iPaD, or phone, assessed by parent completed questionnaire
Tooth Brushing (Caries/Behavioral) | 18 months of age (final follow-up [T2])
  Frequency of parent wiping/brushing teeth, assessed by parent completed questionnaire
Dental Visits (Caries/Behavioral) | 18 months of age (final follow-up [T2])
  Number of dental visits (child), assessed by parent completed questionnaire
Visible Caries | 18 months of age (T2).
  Any visible caries by intra-oral camera (yes/No)
Caries Severity | 18 months of age (T2)
  dfs index
Weight-for-length | 18 months of age (T2)
  BMI-for-age Z scores, standardized for sex and actual age at measurement at the baseline (T0), T1 (12 m.) and T2 (18 m.) interviews. We will categorize children as "overweight" and "obese" if their BMI-for-age Z-scores exceed +2 and +3, respectively, as recommended by the WHO
Change in Weight Velocity Z Scores | see above
  Weight velocity Z scores: for each 6 month period: 6 m.>12 m. 12 m.>18m

CONTACTS AND LOCATIONS:
Overall Officials: Alison Karasz, Principal Investigator — Albert Einstein College of Medicine
Locations (8):
- United States (8):
  - Healthy Kids Pediatric Group, East Windsor, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Smart Medical Care, Jamaica, New York
  - Dr. Masub's Medical and Dental Office, Queens, New York
  - Morris Heights Health Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Group, The Bronx, New York
  - North Central Bronx Hospital, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karasz A, Bonuck K. Reducing pediatric caries and obesity risk in South Asian immigrants: randomized controlled trial of common health/risk factor approach. BMC Public Health. 2018 May 31;18(1):680. doi: 10.1186/s12889-018-5317-9. PMID 29855352